CLINICAL TRIAL: NCT05195723
Title: A Phase 1a, First-in-Human, Randomized, Double-Blind, Placebo-Controlled, Overlapping Single and Multiple Ascending Dose Escalation Study of WP1122 to Establish Maximum Tolerated Dose and Evaluate Pharmacokinetics
Brief Title: Study to Assess the Safety and Pharmacokinetics of WP1122 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Moleculin Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MB-301
Record Dates: First submitted 2021-11-29; First posted 2022-01-19 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — 3,6-di-O-acetyl-2-deoxy-D-glucopyranose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WP1122 (Experimental): Each study group consists of 10 volunteers randomized in a 4:1 ratio to receive WP1122 or placebo. In the first part of the study (Single Ascending Dose [SAD]) in each group (up to 4), 8 volunteers will receive WP1122 and 2 volunteers will receive placebo, one time orally. A total of up to 40 volunteers will be enrolled into the SAD portion of the study.
  The second part of the study (Multiple Ascending Dose [MAD]) will begin when the third group in the SAD part of the study has completed dosing. In this part of the study (MAD) in each group (up to 4), 8 volunteers will receive WP1122 and 2 volunteers will receive placebo, 2 times per day (12 hours apart) orally for 7 days. A total of up to 40 volunteers will be enrolled into the MAD portion of the study.
  Up to 80 volunteers will be enrolled into the study entirely.
  Interventions: Drug: WP1122
- Placebo (Placebo Comparator): Each study group consists of 10 volunteers randomized in a 4:1 ratio to receive WP1122 or placebo. In the first part of the study (Single Ascending Dose [SAD]) in each group (up to 4), 8 volunteers will receive WP1122 and 2 volunteers will receive placebo, one time orally. A total of up to 40 volunteers will be enrolled into the SAD portion of the study.
  The second part of the study (Multiple Ascending Dose [MAD]) will begin when the third group in the SAD part of the study has completed dosing. In this part of the study (MAD) in each group (up to 4), 8 volunteers will receive WP1122 and 2 volunteers will receive placebo, 2 times per day (12 hours apart) orally for 7 days. A total of up to 40 volunteers will be enrolled into the MAD portion of the study.
  Up to 80 volunteers will be enrolled into the study entirely.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: WP1122 — Oral solution
  Arms: WP1122
Drug: Placebo — Oral solution
  Arms: Placebo

SUMMARY:
This study in healthy human volunteers will investigate the effects of a single dose (SAD) and multiple days of dosing (MAD) of WP1122 administered as an oral (PO) solution. Dose escalation will take place in sequential SAD cohorts, and MAD will start as soon as SAD has completed at least 3 dosing cohorts in which WP1122 is found to be safe and well-tolerated. This study in healthy volunteers will explore safety and PK, and subsequent clinical development will be in patients infected with SARS CoV-2 in the setting of continued safety and favorable risk/benefit.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form;
2. Subject is able to understand and comply with protocol requirements, instructions, and protocol-stated restrictions and is likely to complete the study as planned;
3. Male or female, aged 18 to 55 years (inclusive) at the time of signing the informed consent form (ICF);
4. Subject must be willing to undergo COVID-19 testing per clinical pharmacology unit /Phase 1 clinic guidelines;
5. Subject must complete full COVID-19 vaccination course at least 2 weeks prior to study drug administration;
6. Minimum body weight of ≥50 kg (110 lbs) for men and ≥45 kg (99 lbs) for women. Maximum body weight of ≤100 kg (220 lbs). Body Mass Index from 18 to 30 kg/m2 (values rounded to the nearest 10th of a unit);
7. Healthy as determined by a responsible and experienced physician, based on a medical evaluation, including medical history, physical examination, laboratory tests, and ECG:

   1. No evidence of clinically significant cardiac, pulmonary, hepatic, biliary, gastrointestinal, or renal disorders, or cancer within the past 5 years (except localized or in situ cancer of the skin);
   2. Aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase, bilirubin, and creatinine lower than or equal to the ULN. Abnormal values can be repeated once at the discretion of the Investigator or designee;
   3. White blood cell count (including differential), hemoglobin and platelets must be above the lower limit of normal, and if above the ULN, must not be clinically significant in the opinion of the Investigator. A subject with laboratory values outside the reference range may be included at the Investigator's discretion if it is considered clinically insignificant, unlikely to introduce additional risk factors and, in their opinion, does not interfere with study procedures;
8. Women of childbearing potential (WOCBP*) must use a highly effective form of birth control (confirmed by the Investigator). Rhythm methods will not be considered as a highly effective method of birth control. Highly effective forms of birth control include:

   1. Abstinence;
   2. Vasectomized partner (provided that the partner is the sole sexual partner of WOCBP and that the vasectomized partner has received medical assessment of the surgical success);
   3. Oral, intravaginal, or transdermal combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation;
   4. Oral, injectable, or implantable progestogen-only hormone contraception associated with inhibition of ovulation;
   5. Any effective intrauterine device/levonorgestrel intrauterine system;
   6. Female sterilization by tubal occlusion;
   7. WOCBP must agree to use a highly effective method of birth control, as defined above, from the time of signing the ICF, throughout the study duration and until 30 days after the last dose of study drug. Volunteers must have a negative serum pregnancy test result at screening; *WOCBP are defined as women who are NOT permanently sterilized (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy), and who are NOT post-menopausal. Women will be considered post-menopausal if they have been amenorrhoeic for at least 12 months without an alternative medical cause and follicle stimulating hormone (FSH) > 40 IU/mL.
9. Non-vasectomized male volunteers must use an adequate method of contraception (condom with spermicide) from signing the ICF throughout the study duration and until 30 days after the last dose of study drug. Male volunteers must not donate sperm from time of signing the ICF until at least 30 days after the last dose of the study drug.

Exclusion Criteria:

1. Women who are pregnant, breastfeeding or intending to become pregnant, or men intending to father children within the projected duration of the trial from screening until 14 days following last dose;
2. Currently participating in or has participated in a study with an investigational product (IP) within 30 days or 5 half-lives, whichever is longer, preceding Day -1;
3. Due to the current pandemic:

   1. Evidence of current SARS-CoV-2 infection (COVID-19) based on testing at screening;
   2. Documented prior COVID-19 infection in the last 6 months;
   3. Prior COVID 19 infection with ongoing sequelae (i.e., long-hauler COVID), or history of COVID-19 infection requiring an intensive care unit stay or mechanical ventilation;
4. Current or history of the following medical conditions:

   1. Respiratory disease requiring current medical intervention;
   2. Hypersensitivity or severe allergic reactions to vaccines or drugs;
   3. Diagnosis of diabetes mellitus or history of hypo- or hyperglycemia;
   4. Clinically relevant hypertension;
   5. History or active diagnosis of renal disease secondary to diabetes, hypertension, vascular disease;
   6. History of bleeding diathesis or coagulopathy;
   7. Cardiovascular diseases:

   i) QTcF ≥430 msec; History or family history of clinically significant or unstable ECG abnormalities (e.g., prolonged QT syndrome [torsade de pointes] or arrhythmias, including QT prolongation due to medical treatment), sudden cardiac death at a young age, or current use of a QT prolonging drug ii) Angina; iii) Congestive heart failure; iv) Myocardial infarction within the previous 6 months; v) Diastolic dysfunction; vi) Coronary artery disease; h. Malignancy within 5 years of screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy that in the opinion of the Investigator, with concurrence with the Sponsor's Medical Monitor, is considered cured with minimal risk of recurrence);
5. Immunosuppression as a result of underlying illness or treatment including:

   1. Primary immunodeficiencies;
   2. Long-term use (≥7 days) of oral or parenteral glucocorticoids;
   3. Current or anticipated use of disease-modifying doses of antirheumatic drugs and biologic disease-modifying drugs, and no use of such drugs within the last 12 months;
   4. History of solid organ or bone marrow transplantation;
   5. Prior history of other clinically significant immunosuppressive or clinically diagnosed autoimmune diseases;
6. History of substance or alcohol abuse and positive urine drug testing at screening. Subjects with a history of substance or alcohol abuse and negative urine drug testing at screening can be enrolled in study based on the Investigator's discretion;
7. Any physical examination findings and/or history of any illness that, in the opinion of the study Investigator, might confound the results of the study or pose an additional risk to the patient by their participation in the study;
8. Functional disorders of the gastrointestinal (GI) tract and/or surgical procedures that have been conducted (e.g. bariatric surgery, cholecystectomy) which could preclude the ability to adequately allow for effective absorption, distribution, metabolism, or excretion of the drug;
9. Diagnostic Assessments:

   1. A positive test pre-study for hepatitis C antibody, Hepatitis B surface antigen (HbsAg), or human immunodeficiency virus (HIV) antibody;
   2. Hemoglobin A1c ≥ULN;
   3. Serum creatinine greater than or equal to ULN;
   4. Estimated glomerular filtration rate <90 mL/minute as calculated by the chronic kidney disease CKD-EPI formula:

      GFR = 141 * min(Scr/κ,1)α * max(Scr/κ,1) -1.209 * 0.993Age * 1.018 [if female] * 1.159 [if black]
   5. Albumin to creatinine ratio (ACR) ≥0.03 mg/mg. In the event of an ACR above this threshold, eligibility must be confirmed by a second measurement;
   6. Qualitative urinalysis test for blood, or glucose in urine. In the event of a positive test, the test will be repeated once, and if negative, the subject will be considered eligible;
   7. A positive pre-study drug screen or unwilling to refrain from use of the illicit drugs and adhere to other protocol-stated restrictions while participating in the study, including follow-up.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
Safety in Single Ascending Dose (SAD) | 5 weeks
  To investigate the safety and tolerability of escalating doses of WP1122 administered as a single PO dose in sequential cohorts of healthy volunteers and to determine the MTD
Safety in Multiple Ascending Dose (MAD) | 10 weeks
  To investigate the safety and tolerability of 7 days of escalating doses of WP1122 administered q12h PO in sequential cohorts of healthy volunteers and to determine the recommended dose for a Phase 2 trial in patients with COVID-19 (RP2D).

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) in Single Ascending Dose | 5 weeks
  To examine the activity of WP1122 in the body following a single PO dose of WP1122.
Maximum Plasma Concentration (Cmax) in Multiple Ascending Dose | 10 weeks
  To examine the activity of WP1122 in the body following 7 days of q12h PO dosing.

CONTACTS AND LOCATIONS:
Locations (1):
- Medicines Evaluation Unit, Manchester, United Kingdom